CLINICAL TRIAL: NCT01750255
Title: Effect of Pharmaceutical Care in Patients With Bipolar I Disorder at St John of God Clinic. Randomized Trial.
Brief Title: Effect of Pharmaceutical Care in Patients With Bipolar I Disorder (BD I)
Acronym: EMDADER-TABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Humax Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Pedro Amariles, Pharmacy Doctor. Dean of Pharmacy Faculty., Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EMDADER-TABI-20111108
Record Dates: First submitted 2012-08-06; First posted 2012-12-17 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Bipolar Disorder
Keywords: Pharmaceutical care; Pharmacotherapy follow-up; Bipolar disorder; Pharmacy services
MeSH Terms: conditions — Bipolar Disorder | interventions — Pharmaceutical Services; Educational Status; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The control group will receive the usual care and verbal and written information and education about mental health and bipolar disorder for patients and their families. The written material is a brochure designed for this purpose, which focused on the goals and importance of adherence with pharmacological and nonpharmacological interventions to achieve treatment goals. Patients met again with the pharmacist every three months during one year. At each appointment will assess of parameters of efficacy and safety. Quality of life, adherence to treatment, the severity of depressive symptoms in individuals, Symptoms of Mania, the psychiatrist rated patient impairment.
  Interventions: Other: Education
- Pharmaceutical Care (Active Comparator): Pharmaceutical care will be provided according to Dader Method for pharmaceutical care and will be carried out in collaboration with patients and physicians.The time between admission to the group and 20 days,the pharmacist will enhance the information related to treatment adherence and investigate by certain criteria to make an approach to the effectiveness and safety of treatment, through phone calls(weeks 1,3, 4-6) and a home visit(week 2). Pharmacist will call the patient weekly in order to increase adherence. At each appointment will assess of parameters of efficacy (Depression- Mania Rating Scale, Clinical Global Assessment Scale,Quality of life, adherence to treatment.
  Interventions: Other: Pharmaceutical Care

INTERVENTIONS:
Other: Pharmaceutical Care — Pharmaceutical care will be provided according to Dader Method for pharmaceutical care and will be carried out in collaboration with patients and physicians.The time between admission to the group and 20 days,the pharmacist will enhance the information related to treatment adherence and investigate by criteria to make an approach to the effectiveness and safety of treatment, through phone calls(weeks 1,3, 4-6) and a home visit(week 2). Pharmacist will call the patient weekly in order to increase adherence. At each appointment will assess of parameters of efficacy; Depression and Mania Rating Scale, Clinical Global Assessment Scale, Quality of life and adherence to treatment
  Other Names: Pharmacotherapy follow-up; Dader Method for pharmaceutical care
  Arms: Pharmaceutical Care
Other: Education — The control group will receive the usual care and verbal and written information and education about mental health and bipolar disorder for patients and their families. The written material is a brochure designed for this purpose, which focused on the goals and importance of adherence with pharmacological and nonpharmacological interventions to achieve treatment goals. Patients met again with the pharmacist every three months during one year. At each appointment will assess of parameters of efficacy and safety. Quality of life (Sf - 36 test), adherence to treatment, the severity of depressive symptoms in individuals, Symptoms of Mania, the psychiatrist rated patient impairment.
  Other Names: Promotion of health; Disease prevention; Psycho-education
  Arms: Control

SUMMARY:
This project aims, through pharmaceutical care in patients with Bipolar I Disorder, improve compliance and adherence rate, associated with greater effectiveness and safety of drug therapy to help achieve therapeutic goals, and finally to improving the quality of life of patients.

DETAILED DESCRIPTION:
The objective of the present study was to assess the effectiveness of the Dader Method for pharmaceutical care in the reduction of the use of health care services and the increase in the effectiveness and safety of treatment in patients with Bipolar I Disorder who are discharged or referred for outpatient clinic St John of God-La Ceja. Primary objective: To assess the effectiveness of the Dader method for pharmaceutical care on achieving in reducing the number of hospital readmissions, in the increase of the effectiveness and safety of treatment in patients discharged from the Clinic of Saint John of God -La Ceja - Antioquia with bipolar disorder.

A randomized controlled trial. 200 patients will be randomized to group of control or intervention. Post-randomisation, patients will be required to attend the clinic routinely every 3 months during one year. Every 3 months will be evaluated on the criteria of effectiveness and safety of the treatment. Intervention's group will be following through pharmaceutical care. In the development of the study will be a record of the use of health care services (rehospitalizations, care emergency and outpatient, additional to those scheduled).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Bipolar I Disorder
* Have been discharged from the Clinic of Saint John of God -La Ceja-
* Have been resulting from external consultation (outpatient) of the Clinic of Saint John of God -La Ceja-
* Male and female patients aged between 18 and 65 years
* Living in Medellin or any of the following eastern municipalities in the department of Antioquia.

Exclusion Criteria:

* Patients with first episode of manic type, schizoaffective disorder, bipolar disorder II, cyclothymia and other bipolar spectrum disorders, personality disorders that seem bipolar disorder, sociopathic disorder.
* Epilepsy
* Patients unable to comply with the protocol requirements, including severe alcohol and drug use.
* Patients with diagnostic uncertainty.
* Pregnancy or breastfeeding
* Infection with the human immunodeficiency virus (HIV).
* Chronic decompensate disease (no significant diseases): blood pressure values above 180/110 mmHg, total cholesterol above 300 mg / dL, low density cholesterol greater than 160 mmHg, hemoglobin A1c greater than 9%, lower oxygen saturation 90%.
* Mental retardation, presence of any cognitive impairment that prevents understands and signs informed consent.
* Refusal to sign informed consent (Consent must be obtained before any study-related procedures are conducted).
* Illiteracy.
* Patients in electroconvulsive therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salazar, cDr., Study Chair — Universidad de Antioquia; Pedro J Amariles, Dr., Principal Investigator — Universidad de Antioquia; Dora M Benjumea, Dr, Study Chair — Universidad de Antioquia; Luis F Rodriguez, Dr, Study Chair — Clínica San Juan de Dios; Francisco J Gutierrez, Dr, Study Chair — Universidad de Antioquia
Locations (1):
- Clínica San Juan de Dios, La Ceja, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salazar-Ospina A, Amariles P, Benjumea DM, Gutierrez F, Faus MJ, Rodriguez LF. Effectiveness of the Dader Method for pharmaceutical care in patients with bipolar I disorder: EMDADER-TAB: study protocol for a randomized controlled trial. Trials. 2014 May 20;15:174. doi: 10.1186/1745-6215-15-174. PMID 24885673
- [Derived] Salazar-Ospina A, Amariles P, Hincapie-Garcia JA, Gonzalez-Avendano S, Benjumea DM, Faus MJ, Rodriguez LF. Effectiveness of the Dader Method for Pharmaceutical Care on Patients with Bipolar I Disorder: Results from the EMDADER-TAB Study. J Manag Care Spec Pharm. 2017 Jan;23(1):74-84. doi: 10.18553/jmcp.2017.23.1.74. PMID 28025928

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Usual Care (Routine Dispensing), Verbal and Written: Because there is no blinding, there is no 'placebo' treatment. Patients who meet the inclusion criteria will be informed about the study and they will be registered after their signed authorization. The control group (patients and their families) will receive usual care as well as verbal and written information provided by the pharmacist (routine dispensing, including oral counseling regarding drugs). The written material is about mental health (MH) and BD, with information focusing on the importance of adhering to pharmacological and non-pharmacological interventions to achieve treatment goals. Randomization will take place during week zero (baseline) and patients will meet again with the pharmacist every three months (3, 6, 9, and 12 months). At each appointment, variables related to the primary (number of hospitalizations, emergency service consultations, unscheduled outpatient visits) and secondary outcomes (effectiveness, safety, adherence, and quality of life) will be assessed.
- Intervention Group: the Dader Method for Pharmaceutical Care: The Dader Method for pharmaceutical care is a systematic process developed by the Research Group of Pharmaceutical Care at the University of Granada, Spain [16]. The intervention is based on the use of pharmacotherapy records, evaluation of an assessment form that includes BD-I and the drugs used to treat this medical problem, and their assessment on a specific date. This assessment is used to identify: (1) any potential or actual patient health outcomes that are not consistent with the objectives of pharmacotherapy and are associated with the use of medicines (negative outcomes associated with medication (NOM)); and (2) situations in which the use of medicines caused or may cause the appearance of a NOM (drug-related problems (DRP)) [14]. Once the relevant problems are identified, the necessary interventions to patients or to physicians are carried out to solve the identified NOM and are followed by a subsequent assessment of the achieved outcomes.
Period: Overall Study
Arm/Group | Control: Usual Care (Routine Dispensing), Verbal and Written | Intervention Group: the Dader Method for Pharmaceutical Care
Started | 49 | 43
Completed | 43 | 38
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Control: There is no "placebo" treatment, and after randomization, patients were informed of their group assignments. The control group will receive the usual care and verbal and written information and education about mental health and bipolar disorder for patients and their families. The written material is a brochure designed for this purpose, which focused on the goals and importance of adherence with pharmacological and nonpharmacological interventions to achieve treatment goals. Patients met again with the pharmacist every three months during one year. At each appointment will assess of parameters of efficacy and safety. Quality of life, adherence to treatment, the severity of depressive symptoms in individuals, Symptoms of Mania, the psychiatrist rated patient impairment.
  Education: The control group will receive the usual care and verbal and written information and education about mental health and bipolar disorder for patients and their families.
- Pharmaceutical Care: Patients and families will be provided with verbal and written information and education about mental health and bipolar disorder. Pharmaceutical care will be provided according to Dader Method for pharmaceutical care and will be carried out in collaboration with patients and physicians.The time between admission to the group and 20 days,the pharmacist will enhance the information related to treatment adherence and investigate by certain criteria to make an approach to the effectiveness and safety of treatment, through phone calls(weeks 1,3, 4-6) and a home visit(week 2). Pharmacist will call the patient weekly in order to increase adherence. At each appointment will assess of parameters of efficacy (Depression- Mania Rating Scale, Clinical Global Assessment Scale,Quality of life, adherence to treatment. Pharmaceutical Care: Patients and their families will be provided with verbal and written information and education about mental health and bipolar disorder.
- Total: Total of all reporting groups
Arm/Group | Control | Pharmaceutical Care | Total
Number analyzed (Participants) | 49 | 43 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 43 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.8) | 41.9 (9.9) | 42.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Colombia | 49 | 43 | 92

OUTCOME MEASURES:

1. Primary Outcome: To Reduce the Use of Health Care Services by Quantifying the Number of Hospitalizations
Time Frame: 1 year
Measure: Number; unit: Hospitalizations
Arm/Group | Control | Pharmaceutical Care
Number analyzed (Participants) | 49 | 43
Hospitalizations | 12 | 1

2. Primary Outcome: To Reduce the Use of Health Care Services by Quantifying the Number of Emergency Service Consultations
Time Frame: 1 year
Measure: Number; unit: Emergency Service Consultations
Groups:
- Intervention: Pharmaceutical care will be provided according to Dader Method for pharmaceutical care and will be carried out in collaboration with patients and physicians.The time between admission to the group and 20 days,the pharmacist will enhance the information related to treatment adherence and investigate by certain criteria to make an approach to the effectiveness and safety of treatment, through phone calls(weeks 1,3, 4-6) and a home visit(week 2). Pharmacist will call the patient weekly in order to increase adherence. At each appointment will assess of parameters of efficacy (Depression- Mania Rating Scale, Clinical Global Assessment Scale,Quality of life, adherence to treatment.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 49 | 43
Emergency Service Consultations | 23 | 4

3. Primary Outcome: To Reduce the Use of Health Care Services by Quantifying the Number of Unscheduled Outpatient Visits
Time Frame: 1 year
Measure: Number; unit: Outpatient-unscheduled visits
Arm/Group | Control | Intervention
Number analyzed (Participants) | 49 | 43
Outpatient-unscheduled visits | 3 | 12

4. Secondary Outcome: Quality of Life
Description: The Short Form-36 Health Survey (SF-36): It is a questionnaire to measure quality of life, exploring the physical and mental health. Contains 36 topics that explore 8 dimensions of health: physical function; social function; limitations of the role: physical problems; limitations of the role: emotional problems; mental health; vitality; pain and general health perception. Each of the 8 dimensions of the SF-36 scores range between 0 and 100 values. 100 being a result indicating optimal health and 0 would reflect in a very bad state of health. The questionnaire allows the calculation of 2 scores summary, physical component summary (PCS) and mental (MCS), by combining each dimension scores
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Mental health summary score
Arm/Group | Control | Pharmaceutical Care
Number analyzed (Participants) | 49 | 43
Mental health summary score | 83 (22.6) | 89.7 (16.9)

5. Secondary Outcome: Adherence to Treatment
Description: Total percentage of adherence by treatment group
Time Frame: 1 year
Population: Total percentage of adherence by treatment group
Measure: Number; unit: Medication adherence percentage
Arm/Group | Control | Intervention
Number analyzed (Participants) | 49 | 43
Medication adherence percentage | 74.4 | 86.8

6. Secondary Outcome: Clinical Global Impression for Bipolar Modified, CGI-BP-M.
Description: The modified version of the Clinical Global Impression for Bipolar Disorder (CGI-BP-M) a condensed version of the CGI-BP, which is also an adaptation of the CGI for bipolar patients. The CGI-BP-M, is a scale for the assessment of manic, hypomanic, depressive or mixed symptoms, and long-term outcome of bipolar disorder. Assesses the current gravity, the short and long term of the disease course. It consists of three subscales, composed of a single item, evaluating the severity of the acute symptoms of depression, mania and disease in general (refers to the longitudinal disease severity). It has a Likert intensity scale of 7 degrees of freedom ( 1 normal, 7 very severe).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Clinical Global Impression
Arm/Group | Control | Intervention
Number analyzed (Participants) | 49 | 43
Clinical Global Impression | 1.6 (0.7) | 1.3 (0.6)

7. Secondary Outcome: Mania
Time Frame: 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Depression
Description: To assess depressive symptoms, will be used the the Hamilton Depression Rating Scale. [Time Frame: At 3, 6, 9 and 12 months]using hamilton depression scale
Time Frame: 1 year
Reporting Status: Not Posted

9. Secondary Outcome: Necessity, Effectiveness and Security Problems Associated With Pharmacotherapy
Description: Necessity problems of pharmacotherapy are related to the following two questions: 1) The patient has a health problem associated with not receiving a medication you need? 2) The patient has a health problem associated with getting a medicine that does not need. The safety of the pharmacotherapy will be measured by the safety profile of drugs and serum concentrations of drugs. The effectiveness of the pharmacotherapy will be measured by Hamilton Rating Scale for Depression, Clinical Global Impressions (CGI), Young Mania Rating Scale.
Time Frame: 1 year
Reporting Status: Not Posted

10. Secondary Outcome: Preventable Causes of Problems of Effectiveness and Safety of Pharmacotherapy
Description: Quantify the preventable causes of problems of effectiveness and safety of pharmacotherapy. Quantify the process problems like a drug availability problems, problems in prescribing, dispensing problems, administration and use, quality problem.[Time Frame: At 3, 6, 9 and 12 months]
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Control: The control group will receive the usual care and verbal and written information and education about mental health and bipolar disorder for patients and their families. The written material is a brochure designed for this purpose, which focused on the goals and importance of adherence with pharmacological and nonpharmacological interventions to achieve treatment goals. Patients met again with the pharmacist every three months during one year. At each appointment will assess of parameters of efficacy and safety. Quality of life, adherence to treatment, the severity of depressive symptoms in individuals, Symptoms of Mania, the psychiatrist rated patient impairment.
  Education: The control group will receive the usual care and verbal and written information and education about mental health and bipolar disorder for patients and their families. The written material is a brochure d
- Pharmaceutical Care: Patients and families will be provided with verbal and written information and education about mental health and bipolar disorder. Pharmaceutical care will be provided according to Dader Method for pharmaceutical care and will be carried out in collaboration with patients and physicians.The time between admission to the group and 20 days,the pharmacist will enhance the information related to treatment adherence and investigate by certain criteria to make an approach to the effectiveness and safety of treatment, through phone calls(weeks 1,3, 4-6) and a home visit(week 2). Pharmacist will call the patient weekly in order to increase adherence. At each appointment will assess of parameters of efficacy (Depression- Mania Rating Scale, Clinical Global Assessment Scale,Quality of life, adherence to treatment.
Arm/Group | Control | Pharmaceutical Care
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/43
Other Adverse Events (participants affected / at risk) | 0/49 | 0/43

LIMITATIONS AND CAVEATS:
There was no "placebo" treatment, the study patients were not blinded to treatment assignment and both groups (were seen by the same pharmacist, who was responsible for collecting the measurements).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No